CLINICAL TRIAL: NCT04909164
Title: The Pragmatic Clinical Trial to Elucidate Optimal Target Population of Immunotherapy From Real-world Lung Cancer Patients
Brief Title: The Prospective Non-randomized Case-control Study From Real-world Lung Cancer Patients
Acronym: OPTIMUS
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-02-015
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 2nd-line Immunotherapy group: Patients receiving reimbursed immunotherapy as a second-line therapy (in case of targeted therapy, patients receiving immunotherapy after targeted therapy-platinum-based chemotherapy) Drugs name : Pembrolizumab, Atezolizumab ,Nivolumab
  Interventions: Drug: Immunnotherapy group
- 2nd-line Cytotoxic chemotherapy group: Patients receiving reimbursed cytotoxic chemotherapy as second-line therapy after failure of platinum-based chemotherapy Drugs name : Docetaxel
  Interventions: Drug: Immunnotherapy group
- 1st-line Immunotherapy group: First- line Control Arm: Retrospective hisrotical data of 680 cases to be collected Drugs name :Pembrolizumab only Pembrolizumab + Pemetrexed + Carboplatin Pembrolizumab + Paclitaxel + Carboplatin
  Interventions: Drug: Immunnotherapy group
- 1st- line Cytotoxic chemotherapy group(retrospective): ⦁ Retrospective: In addition to the prospective data, retrospective data will be collected from medical records of 680 patients (or more) who had records of receiving cytotoxic chemotherapy between January 1, 2017, and December 31, 2018 (1:1 comparison between the immunotherapy arm and the chemotherapy arm). If the patient did not die within the first 12 months after diagnosis, available follow-up data of at least 12 months will be collected from the medical records of the participating institution.
  Drugs name :
  Pemetrexed + Cisplatin/Carboplatin Gemcitabine + Cisplatin/Carboplatin
  Interventions: Drug: Immunnotherapy group

INTERVENTIONS:
Drug: Immunnotherapy group — Eligible patients are those who receive reimbursed immunotherapy or cytotoxic chemotherapy after failure of platinum-based chemotherapy per current health insurance reimbursement criteria.
  Other Names: Cytotoxic chemotherapy group

SUMMARY:
The pragmatic clinical trial to elucidate optimal target population of immunotherapy from real-world lung cancer patients

DETAILED DESCRIPTION:
Eligible patients are those who receive reimbursed immunotherapy or cytotoxic chemotherapy after failure of platinum-based chemotherapy per current health insurance reimbursement criteria. This study will not provide any additional intervention to patients, but they will receive all treatments available per standard of care at each institution. If the reimbursement criteria change or expand (to include the immunotherapy as the first-line therapy) in the future, patients who get to receive immunotherapy or cytotoxic chemotherapy according to the revised and expanded reimbursement criteria will be enrolled as well.

Because immunotherapy was superior to the existing cytotoxic chemotherapy in terms of survival and AEs in previous large-scale prospective studies, immunotherapy has been preferred than cytotoxic chemotherapy after failure of platinum-based chemotherapy in real-world clinical settings. In addition, pembrolizumab and nivolumab are reimbursed according to PD-L1 expression levels, but atezolizumab is reimbursed for all patients regardless of PD-L1 expression levels and thus is available for reimbursed prescription for practically every patient. These three agents showed almost no difference in their clinical effectiveness in previous prospective global studies. However, cytotoxic chemotherapy is selected over immunotherapy in some patients, and they will be assigned to the control group.

Based on the patient's symptoms and the physician's clinical judgment, cytotoxic therapy can be selected as a second-line therapy in clinical settings if the patient has an extensive lesion that requires inducing a rapid response or has experienced a disease progression centered on bone or liver metastases, which are known to respond only marginally to immunotherapy.

ELIGIBILITY:
7-1 Inclusion criteria 7-1-1 Immunotherapy arm (prospective data collection)

* Male and female patients aged 19 years and above
* Patients with histologically confirmed NSCLC
* Patients on palliative therapy for recurrence after surgery or de novo advanced and metastatic disease
* Patients receiving reimbursed immunotherapy as second-line therapy (in case of targeted therapy, patients receiving immunotherapy after targeted therapy-platinum-based chemotherapy) or as reimbursed first-line therapy
* Patients who provided written informed consent for the study (including the secondary use of the study data and sharing with third parties) 7-1-2 Cytotoxic chemotherapy arm (prospective/retrospective data collection)
* Male and female patients aged 19 years and above
* Patients with histologically confirmed NSCLC
* Patients on palliative therapy for recurrence after surgery or de novo advanced and metastatic disease
* Prospective: Patients receiving reimbursed cytotoxic chemotherapy as second-line therapy after failure of platinum-based chemotherapy
* Retrospective: In addition to the prospective data, retrospective data will be collected from medical records of 680 patients (or more) who had records of receiving cytotoxic chemotherapy between January 1, 2017, and December 31, 2018 (1:1 comparison between the immunotherapy arm and the chemotherapy arm). If the patient did not die within the first 12 months after diagnosis, available follow-up data of at least 12 months will be collected from the medical records of the participating institution.Patients who provided written informed consent for the study (including the secondary use of the study data and sharing with third parties) 7-2 Exclusion criteria 7-2-1 Immunochemotherapy arm
* Patients receiving immunotherapy without reimbursement
* Patients who do not provide consent to the study 7-2-2 Cytotoxic chemotherapy arm
* Patients receiving cytotoxic chemotherapy without reimbursement
* Patients who do not provide consent to the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: real-world lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 3 years
  The time from first dose to disease progression or death from any cause
Overall-survival | Up to 3 years
  The time from first dose to death from any cause

SECONDARY OUTCOMES:
Response rate | Up to 3 years
  The proportion of patients showing complete or partial response as determined by RECIST v1.1
Disease control rate | Up to 3 years
  The proportion or patients showing complete or partial response or stable disease as determined by RECIST v1.1.
Duration of response | Up to 3 years
  The duration of response in patients showing complete or partial response
Hyper-progression | Up to 3 years
  The proportion of patients showing hyper-progression after prior treatment according to the criterion for hyper-progression, their survival rate, and predictors of survival

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, M.D, Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No